CLINICAL TRIAL: NCT01088282
Title: Visual Function, Non-dependence on Glasses and Global Economic Cost in Patients Undergoing Lens Surgery With ReSTOR® Multifocal Aspheric Iol Implants
Brief Title: Visual and Economic Profits of ReSTOR® Multifocal Intraocular Lenses (IOL) on Public Health Patients in Spain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Josep Torras MD, Hospital Clinic Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECICOFPALIORES09
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-02

CONDITIONS: Presbyopia
Keywords: Diffractive multifocal IOL
MeSH Terms: conditions — Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implantation of difractive multifocal IOL (Active Comparator)
  Interventions: Procedure: Cataract surgery
- Implantation of monofocal IOL (Sham Comparator)
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Implantation of multifocal or monofocal IOL
  Other Names: SN6AD1 (Alcon labs, Fotworth, Texas) in active comparator; SN60WF (Alcon labs, Fotworth, Texas) in sham comparator

SUMMARY:
Surgical correction of presbyopia is possible via the implantation of multifocal intraocular lenses after removal of the crystalline lens. The cost of these implants is approximately 6 times higher than the conventional monofocal implants routinely used in all crystalline surgery for correction of the resulting ametropia. Spectacles for correcting presbyopia, which are necessary after the insertion of monofocal implants, may also have a significant cost.

The proposed trial will involve two randomized groups of patients in need of crystalline/cataract surgery, with monofocal or multifocal lens implants (the same type of lens in both eyes) leaving them emmetropic for distant vision.

The objective is to corroborate with blind-evaluation the effectiveness of multifocal lens implants in obviating the need for glasses to correct presbyopia, to evaluate the benefits of this type of implant, both in global economic terms (adding the cost of the implants to that of corrective glasses where necessary) and in terms of the improved quality of life of the patients, and to confirm the absence of adverse effects.

Findings will be subjected to a statistical quantification.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 50 and over, with fully-established presbyopia, requiring phacoemulsification + IOL as the surgical technique for the removal of their cataracts.
* Their capsular bags should be stable, with keratometric astigmatism equal to or lower than 1 diopter.
* Biometric calculations should indicate an IOL for emmetropy within the common dioptric range for both lenses, i.e. between +6 y +34.

Exclusion Criteria:

* Previous corneal refractive surgery
* Maculopathy, amblyopia or other eye conditions that limit visual power
* Occupations requiring special driving licenses
* Keratometric astigmatism higher than 1 diopter
* Any intraoperative posterior capsular rupture or extracapsular reconversion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Visual function quality (VF-14) | At 1 and 3 months post-intervention

SECONDARY OUTCOMES:
Visual acuity with and without correction | at 1 and 3 months post-intervention
Determine Expense in glasses | at 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Josep Torras, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic. Casa Maternitat, Barcelona, Barcelona
  - Hospital Clinic. Casa maternitat, Barcelona, Barcelona